CLINICAL TRIAL: NCT02612649
Title: Special Drug Use Surveillance of Irribow® Tablets and Irribow® OD Tablets in Female Patients
Brief Title: Special Drug Use Surveillance of Irribow in Female Patients
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: IB0002
Record Dates: First submitted 2015-10-23; First posted 2015-11-24 (Estimated); Last update posted 2024-10-21 (Actual); Status verified 2018-10

CONDITIONS: Diarrhea-predominant Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; YM060; Ramosetron; Survey
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — ramosetron

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ramosetron group: Female patients with diarrhea-predominant irritable bowel syndrome
  Interventions: Drug: Ramosetron

INTERVENTIONS:
Drug: Ramosetron — Oral
  Other Names: YM060; Irribow

SUMMARY:
The purpose of the survey is to evaluate the safety and efficacy of Irribow and Irribow OD Tablets in post-marketing medical practice and to examine the status of treatment compliance.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with diarrhea-predominant irritable bowel syndrome

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female patients with diarrhea-predominant irritable bowel syndrome
Sampling Method: Non-Probability Sample
Enrollment: 793 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Incidences of Adverse Drug Reactions | Up to Week 52

SECONDARY OUTCOMES:
Change from baseline in frequency of bowel movements | Baseline to Week 52
  Frequency of bowel movements is recorded daily
Change from baseline in form of stool | Baseline to Week 52
  Classified based on Bristol Stool Form Scale
Change from baseline in sensation of incomplete bowel evacuation | Baseline to Week 52
  Assessment based on numerical rating scale
Change from baseline in defecation urgency | Baseline to Week 52
Change from baseline in abdominal pain or discomfort | Baseline to Week 52
  Abdominal pain or discomfort assessed based on numerical rating scale
Change from baseline in melena | Baseline to Week 52
Overall improvement | Up to Week 52
  Classified into the three scales (improved, no change or aggravated) or concluded as indeterminable.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (34):
- Japan (34):
  - Numakunai, Iwate
  - Aichi
  - Akita
  - Chiba
  - Fukui
  - Fukuoka
  - Fukushima
  - Gifu
  - Gunma
  - Hiroshima
  - Hyōgo
  - Ibaraki
  - Kagoshima
  - Kanagawa
  - Kumamoto
  - Kyoto
  - Mie
  - Miyagi
  - Miyazaki
  - Nagano
  - Niigata
  - Okayama
  - Okinawa
  - Osaka
  - Ōita
  - Saitama
  - Shiga
  - Shizuoka
  - Tochigi
  - Tokyo
  - Tottori
  - Toyama
  - Yamagata
  - Yamaguchi

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.